CLINICAL TRIAL: NCT06087497
Title: The Z Stitch Early Bed Rest Assessment Study
Acronym: ZEBRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Charles Henrikson, MD, Director Electrophysiology, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00025985
Record Dates: First submitted 2023-10-12; First posted 2023-10-17 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Atrial Fibrillation; Atrial Flutter; Supraventricular Tachycardia; Syncope; Ventricular Tachycardia
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Tachycardia, Supraventricular; Syncope; Tachycardia, Ventricular | interventions — Early Ambulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 hour bedrest (Experimental): One hour of bedrest, elevate head of bed to 30 degrees at 30 minutes, ambulate at 60 minutes, Z stitches out at 4 hours, eligible for discharge (if appropriate) at 4.5 hours.
  Interventions: Other: Early mobilization
- 4 hour bedrest (No Intervention): Four hours of bedrest, elevate head of bed to 30 degrees at 2 hours, Z stitches out at 4 hours, ambulate at 4 hours, eligible for discharge at 4.5 hours.

INTERVENTIONS:
Other: Early mobilization — Z stitch placement is standard of care to achieve vascular hemostasis after EP procedures which is followed by 4 hours of bedrest. In this study, we will compare patient satisfaction and bleeding complications with a shorter bedrest (1 hour instead of 4 hours)
  Arms: 1 hour bedrest

SUMMARY:
The goal of this study is to understand the effects of early mobilization after a Z stitch procedure in patients undergoing certain heart-related treatments. The investigators want to find out if allowing patients to move around sooner after their procedure can improve their satisfaction and potentially lead to earlier discharge from the hospital.

Type of Study: Clinical Trial

Participant Population/Health Conditions: Patients aged 18-99 undergoing specific heart procedures such as atrial fibrillation treatment, atrial flutter treatment, supraventricular tachycardia treatment, diagnostic electrophysiology studies, AV node ablation, or Watchman device placement.

Main Questions:

Does early mobilization (getting up and moving around sooner) after the Z stitch procedure improve patient satisfaction?

Participants will be divided into two groups, and researchers will compare those who have one hour of bedrest with those who have four hours of bedrest after the Z stitch procedure. The investigators want to see if the shorter bedrest period leads to higher patient satisfaction.

DETAILED DESCRIPTION:
The ZEBRA study, or the Z stitch Early Bed Rest Assessment study, aims to assess the impact of early mobilization following Z stitch placement on patient satisfaction and safety in the context of venous vascular access management during Electrophysiology (EP) procedures. The study hypothesizes that allowing patients to move sooner after Z stitch placement will lead to higher patient satisfaction scores without compromising safety. The primary endpoint for evaluation is patient satisfaction, gauged through survey-based scores, while secondary endpoints encompass a range of factors including hematoma development, bleeding-related complications, the use of pain medications, associated healthcare costs, 30-day patient outcomes, actual post-procedure ambulation time, and instances of hospital readmissions or emergency department visits within the initial 30 days post-procedure.

Historically, venous vascular access has been managed by employing direct manual pressure for hemostasis following sheath removal, which necessitates a prolonged period of bed rest for the patient. However, a recent advancement, termed the "Z stitch" method, achieves hemostasis by placing a Z-shaped stitch around the vascular access site, providing continuous pressure and allowing for safer sheath removal without the need for anticoagulation reversal. Despite the effectiveness of the Z stitch, current practice still involves extended bed rest post-procedure. This randomized clinical trial aims to fill the existing knowledge gaps by approaching eligible patients ahead of their procedures or during the consent process. Patients will be randomized 1:1 to two distinct protocols: one involving one hour of bed rest post-procedure, followed by ambulation at 60 minutes and Z stitch removal at 4 hours; and the other entailing 4 hours of bed rest, with Z stitch removal and ambulation at the same 4-hour mark. Compression time at the Z stitch placement will also be stratified based on the sheath size and whether systemic anticoagulation is used. Assessments for groin hematoma and patient satisfaction surveys will be completed prior to discharge, with a 30-day phone follow-up to evaluate longer-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

Presenting for procedure in the EP lab for:

* Atrial fibrillation
* Atrial flutter
* Supraventricular tachycardia
* Diagnostic EP study
* Atrioventricular node ablation
* Watchman device placement

Exclusion Criteria:

* Those who refuse or are unable to consent.
* Cases involving arterial access.
* Cases involving access with a >16Fr sheath (i.e., no leadless pacer patients).
* Patients with a BMI > 40.
* Lead-extraction patients.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | At the time of discharge
  Patient satisfaction will be assessed with a survey prior to discharge.

SECONDARY OUTCOMES:
Complications | 30 days from the procedure
  Rates of hematomas, Other bleeding complications, Other complications, Use of pain medications, Cost, 30 day outcomes, Readmission/ED visit for groin concerns within 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Henrikson, MD, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Oregon Health and Science University, Portland, Oregon
  - Portland VA Medical Center, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) with other researchers